CLINICAL TRIAL: NCT02114008
Title: Residual Gastric Volume in Morbidly Obesa Diabetics. A Comparison of 3 Hour Versus Hour Fasting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cuiaba University (Other)
Responsible Party: Principal Investigator, Gunther Peres Pimenta, MD, PhD, Cuiaba University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 179.017/2012 CEP UFMT
Record Dates: First submitted 2014-04-12; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Obesity; Diabetes; Fasting
Keywords: Gastric emptying.; Residual gastric volume.; Preoperative fasting.; Morbid Obesity.; Diabetes.
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Fasting; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abbreviated fasting (Active Comparator): Patients underwent two endoscopic examinations within two weeks. RGV was measured by aspiration of gastric contentes into a graduated cylinder after traditional after abbreviated fasting (3 hours with 200ml of water containing 25g of 12.5% maltodextrin).
  Interventions: Other: Endoscopic examinations
- Traditional fasting (Active Comparator): Patients underwent two endoscopic examinations within two weeks. RGV was measured by aspiration of gastric contentes into a graduated cylinder after traditional fasting (at least 8 hours before the test).
  Interventions: Other: Endoscopic examinations

INTERVENTIONS:
Other: Endoscopic examinations — Patients underwent two endoscopic examinations within two weeks. RGV was measured by aspiration of gastric contentes into a graduated cylinder after traditional fasting (at least 8 hours before the test) and after abbreviated fasting (3 hours with 200ml of water containing 25g of 12.5% maltodextrin). All patients received both oral and written information about the protocol at the outpatient clinic.

SUMMARY:
To reduce the risk of aspiration for elective procedures, residual gastric volumes (RGV) have traditionally been minimized with overnight fasting. However, prolonged fasting can also have some adverse consequences and has been abandoned for some procedures in several patient populations with the exception of obese and/or diabetic patients. The aim of this study was to assess RGV in morbidly obese diabetic patients after traditional or abbreviated fasting.

DETAILED DESCRIPTION:
Patients underwent two endoscopic examinations within two weeks. RGV was measured by aspiration of gastric contentes into a graduated cylinder after traditional fasting (at least 8 hours before the test) and after abbreviated fasting (3 hours with 200ml of water containing 25g of 12.5% maltodextrin). All patients received both oral and written information about the protocol at the outpatient clinic.

All the endoscopic procedures began at 9 AM, and were performed by the same board-certified endoscopist, JMS, who was blinded as to the duration of the fast. The endoscopies were conducted at Gastroclinica, Cuiaba, MT, in the period from April to June, 2013. Sedation was performed by a board-certified anesthesiologist, who was also blinded as to the duration of the fast. The anesthetic regimem included a intravenous bolus of 2 ml of lidocaine hydrochloride (Astra Zeneca, São Paulo, Brazil) followed by 100 to 150mg of propofol before endoscopy. Digital oximetry was monitored throughout the procedure. Patients were positioned in the lateral recumbent position. A flexible electronic videoendoscope (EG2770K; Pentax Corporation, Tokyo, Japan) of 9 mm in outer diameter was used. The main outcome variable was the RGV measured by the endoscopist after aspiration of gastric residue.

ELIGIBILITY:
Inclusion Criteria: patients between 18 and 55 years of age, of both sexes, with Body Index Mass (BMI) which is equal or greater than 40 Kg/m2, and type II diabetic that were using oral drugs or insulin to control the disease.

-

Exclusion Criteria: patients who were using medications for gastrointestinal symptoms and/or who had prior abdominal operations.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Residual gastric volume (RGV) in morbidly obese diabetics. A comparison of 3 hour versus 8 hour fasting | 3 months
  This was a prospective, randomized, double-blind, and cross-over design in 8 morbidly obese type II diabetics with informed consent. RGV was measured endoscopically after three and eight hour fasts.

CONTACTS AND LOCATIONS:
Overall Officials: Gunther P Pimenta, MD, PhD, Principal Investigator — Cuiaba University
Locations (1):
- Gunther Peres Pimenta, Cuiabá, Mato Grosso, Brazil